CLINICAL TRIAL: NCT02243202
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Safety and Efficacy of the Co-administration of Canagliflozin 300 mg and Phentermine 15 mg Compared With Placebo for the Treatment of Non-diabetic Overweight and Obese Subjects
Brief Title: Effects of Co-administration of Canagliflozin 300 mg and Phentermine 15 mg With Placebo in the Treatment of Non-Diabetic Overweight and Obese Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103086; 28431754OBE2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Canagliflozin; Phentermine; INVOKANA®
MeSH Terms: conditions — Obesity; Overweight | interventions — Canagliflozin; Phentermine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Canagliflozin + Phentermine (Experimental): 300 mg capsule of Canagliflozin along with 15 mg capsule of Phentermine, taken once daily, orally for 26 weeks.
  Interventions: Drug: Canagliflozin; Drug: Phentermine
- Canagliflozin + Placebo (Phentermine) (Experimental): 300 mg capsule of Canagliflozin along with matching placebo to Phentermine, taken once daily, orally for 26 weeks.
  Interventions: Drug: Canagliflozin; Drug: Matching Placebo to Phentermine
- Phentermine + Placebo (Canagliflozin) (Experimental): 15 mg capsule of Phentermine along with matching placebo to Canagliflozin, taken once daily, orally for 26 weeks.
  Interventions: Drug: Phentermine; Drug: Matching Placebo to Canagliflozin
- Placebo (Placebo Comparator): Matching placebo to Canagliflozin and Phentermine, taken once daily, orally for 26 weeks.
  Interventions: Drug: Matching Placebo to Canagliflozin; Drug: Matching Placebo to Phentermine

INTERVENTIONS:
Drug: Canagliflozin — 300 mg capsule, taken once daily, orally for 26 weeks.
  Other Names: INVOKANA
  Arms: Canagliflozin + Phentermine; Canagliflozin + Placebo (Phentermine)
Drug: Phentermine — 15 mg capsule, taken once daily, orally for 26 weeks.
  Arms: Canagliflozin + Phentermine; Phentermine + Placebo (Canagliflozin)
Drug: Matching Placebo to Canagliflozin — Placebo capsules look like canagliflozin but do not contain any active drug, taken once daily, orally for 26 weeks.
  Arms: Phentermine + Placebo (Canagliflozin); Placebo
Drug: Matching Placebo to Phentermine — Placebo capsules look like phentermine but do not contain any active drug, taken once daily, orally for 26 weeks.
  Arms: Canagliflozin + Placebo (Phentermine); Placebo

SUMMARY:
The purpose of this study is to compare the effects of canagliflozin and phentermine to those of placebo to promote on a change in body weight over a 26 week period.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect), parallel-group, multicenter study of the effects of canagliflozin and phentermine co-administration in non-diabetic overweight or obese participants. The study will be conducted for about 33 weeks, approximately 344 participants will be randomly assigned in a 1:1:1:1 ratio to one of the four treatment groups: co-administration of canagliflozin and phentermine, canagliflozin alone, phentermine alone, or placebo. All participants will be also provided with diet and exercise counseling for weight loss (standardized non-pharmacological therapy).

ELIGIBILITY:
Inclusion Criteria:

* Must have BMI >=30 kg/m2 and <50 kg/m2 at screening or BMI >=27 kg/m2 and <50 kg/m2 at screening in the presence of a comorbidity of hypertension and/or dyslipidemia
* Must have stable weight, ie, change of < =5% in the 3 months before screening
* Must agree to utilize a highly effective method of birth control

Exclusion Criteria:

* An established diagnosis of diabetes mellitus
* Has a history of obesity with a known secondary cause (eg, Cushing's disease/syndrome)
* Has a history of hereditary glucose-galactose malabsorption or primary renal glycosuria
* Myocardial infarction, unstable angina, revascularization procedure, or cerebrovascular accident within 12 weeks before screening
* Has an Glycated hemoglobin (HBA1c) greater than or equal (>=) to 65 percent
* An average of 3 seated blood pressure (BP) readings of systolic BP >= 160 mm Hg and/or Diastolic BP >= 100 millimeters of mercury at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (17):
  - Phoenix, Arizona
  - Walnut Creek, California
  - Jacksonville, Florida
  - Meridian, Idaho
  - Evansville, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Milford, Massachusetts
  - Manlius, New York
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Odessa, Texas
  - Norfolk, Virginia
  - Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between screening and randomisation, eligible subjects were included in a 4-week single-blind run-in period in which all subjects were placed on a hypocaloric diet.
Groups:
- Placebo: Participants received placebo tablets orally for 26 weeks.
- Phentermine 15 mg: Participants received phentermine 15 mg over-encapsulated tablets orally for 26 weeks.
- Canagliflozin 300 mg: Participants received canagliflozin 300 mg over-encapsulated tablets orally for 26 weeks.
- Canagliflozin 300 mg/Phentermine 15 mg: Participants received co-administration of canagliflozin 300 mg and phentermine 15 mg orally for 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Started | 82 | 85 | 84 | 84
Treated | 82 | 85 | 84 | 83
Completed | 57 | 60 | 53 | 61
Not Completed | 25 | 25 | 31 | 23
Not completed — Adverse Event | 5 | 6 | 10 | 4
Not completed — Lost to Follow-up | 9 | 9 | 14 | 11
Not completed — Protocol Violation | 3 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 4 | 4
Not completed — Other | 1 | 3 | 1 | 2
Not completed — Randomized but not received treatment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of double-blind study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg | Total
Number analyzed (Participants) | 82 | 85 | 84 | 83 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (11.09) | 46.4 (11.14) | 45.2 (11.02) | 46.3 (12.45) | 45.7 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 68 | 69 | 273
  Male | 15 | 16 | 16 | 14 | 61
Region of Enrollment [Number; unit: participants]
  United States | 82 | 85 | 84 | 83 | 334
Baseline Weight [Mean (Standard Deviation); unit: Kilogram [kg]] | 104.3 (18.16) | 102.8 (17.89) | 103.3 (19.14) | 101.1 (18.07) | 102.9 (18.28)
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter square [kg/m²]] | 38 (5.2) | 37 (5.4) | 37.3 (4.68) | 36.8 (5.36) | 37.3 (5.16)
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury [mmHg]] | 122.5 (13.86) | 123.0 (11.83) | 124.5 (13.01) | 124.8 (12.83) | 123.7 (12.87)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury [mmHg]] | 78.8 (8.43) | 78.1 (9.00) | 80.2 (7.88) | 79.4 (8.21) | 79.1 (8.39)
Baseline Pulse Rate [Mean (Standard Deviation); unit: (BEATS/MIN)] | 73.5 (8.72) | 70.7 (10.09) | 71.5 (9.40) | 72.4 (9.66) | 72.0 (9.50)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at Week 26
Description: The percent change from baseline in body weight at Week 26 was analysed.
Time Frame: Week 26
Population: The modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of double-blind study agent. N=number of participants analysed is the total participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 76 | 76 | 78 | 77
Percent Change | -0.6 (0.6) | -4.1 (0.6) | -1.9 (0.6) | -7.5 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Phentermine 15 mg; Test type: Superiority or Other; p < 0.001, Mixed Model for Repeated Measures; Least Square Mean Difference = -3.5, 95% CI 2-sided [-5.3 to -1.8], Standard Error of Mean 0.9
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.142, Mixed Model for Repeated Measures; Least Square Mean Difference = -1.3, 95% CI 2-sided [-3.1 to 0.4], Standard Error of Mean 0.9
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg/Phentermine 15 mg; Test type: Superiority or Other; p < 0.001, Mixed Model for Repeated Measures; Least Square Mean Difference = -6.9, 95% CI 2-sided [-8.6 to -5.2], Standard Error of Mean 0.9

2. Secondary Outcome: Percentage of Participants With Weight Loss More Than Equal to (>=) 5 Percent at Week 26
Description: Percentage of participants with weight loss >= 5 percent were analysed at week 26.
Time Frame: Week 26
Population: The mITT analysis set included all randomized participants who received at least 1 dose of double-blind study agent. N=number of participants analysed is the total participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 57 | 60 | 56 | 63
percentage of participants | 17.5 | 41.7 | 17.9 | 66.7
Statistical Analysis 1: Comparison: Placebo vs Phentermine 15 mg; Test type: Superiority or Other; p = 0.002, Generalized linear Mixed Model; Odds Ratio (OR) = 4.15, 95% CI 2-sided [1.70 to 10.14]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.825, Generalized linear Mixed Model; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.41 to 3.06]
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg/Phentermine 15 mg; Test type: Superiority or Other; p < 0.001, Generalized linear Mixed Model; Odds Ratio (OR) = 10.20, 95% CI 2-sided [4.15 to 25.05]

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 26
Description: Change from baseline in systolic blood pressure was analysed at week 26.
Time Frame: Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 75 | 76 | 78 | 77
mmHg (millimeters of mercury) | -2.7 (1.3) | -1.4 (1.2) | -3.1 (1.3) | -6.9 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Phentermine 15 mg; Test type: Superiority or Other; p = 0.456, Mixed Model for Repeated Measures; Least Square Mean Difference = 1.3, 95% CI 2-sided [-2.1 to 4.8], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.827, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.4, 95% CI 2-sided [-3.9 to 3.1], Standard Error of Mean 1.8
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg/Phentermine 15 mg; Test type: Superiority or Other; p = 0.015, Mixed Model for Repeated Measures; Least Square Mean Difference = -4.2, 95% CI 2-sided [-7.7 to -0.8], Standard Error of Mean 1.7

4. Secondary Outcome: Absolute Change From Baseline in Body Weight at Week 26
Description: Absolute change from baseline in body weight was analysed at week 26.
Time Frame: Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Kilogram (Kg)
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 76 | 76 | 78 | 77
Kilogram (Kg) | -0.6 (0.6) | -4.1 (0.6) | -1.9 (0.7) | -7.3 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Phentermine 15 mg; Test type: Superiority or Other; p < 0.001, Mixed Model for Repeated Measures; Least Square Mean Difference = -3.5, 95% CI 2-sided [-5.3 to -1.7], Standard Error of Mean 0.9
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.153, Mixed Model for Repeated Measures; Least Square Mean Difference = -1.3, 95% CI 2-sided [-3.1 to 0.5], Standard Error of Mean 0.9
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg/Phentermine 15 mg; Test type: Superiority or Other; p < 0.001, Mixed Model for Repeated Measures; Least Square Mean Difference = -6.7, 95% CI [-8.5 to -4.9], Standard Error of Mean 0.9

5. Other Pre Specified Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Week 26
Description: Change from baseline in diastolic blood pressure (DBP) at week 26.
Time Frame: Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 75 | 76 | 78 | 77
mmHg (millimeters of mercury) | -0.9 (0.9) | 0.1 (0.8) | -1.5 (0.9) | -2.5 (0.8)

6. Other Pre Specified Outcome: Change From Baseline in Pulse Rate at Week 26
Description: Change from baseline in pulse rate at week 26
Time Frame: Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Beats Per Minute (Beats/Min)
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 75 | 76 | 78 | 77
Beats Per Minute (Beats/Min) | -0.7 (1.0) | 4.1 (1.0) | 0.7 (1.0) | 3.5 (0.9)

7. Other Pre Specified Outcome: Percentage of Participants With Weight Loss More Than Equal to (>=) 10 Percent at Week 26
Description: Percentage of participants with weight loss >= 10 percent at week 26.
Time Frame: Week 26
Population: The mITT analysis set included all randomized participants who received at least 1 dose of double-blind study agent.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Number analyzed (Participants) | 82 | 85 | 84 | 83
Percentage of Participants | 8.8 | 8.3 | 5.4 | 34.9

ADVERSE EVENTS:
Time Frame: Up to 33 weeks
Description: Only participants who had TEAE (Treatment-Emergent Adverse Event) in the table (i.e. meeting the pre-specified cut-off percentage) are included in the Total, other (not including serious) adverse events count.
Arm/Group | Placebo | Phentermine 15 mg | Canagliflozin 300 mg | Canagliflozin 300 mg/Phentermine 15 mg
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/85 | 0/84 | 1/83
Other Adverse Events (participants affected / at risk) | 41/82 | 37/85 | 42/84 | 42/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Phentermine 15 mg (N=85) | Canagliflozin 300 mg (N=84) | Canagliflozin 300 mg/Phentermine 15 mg (N=83)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Phentermine 15 mg (N=85) | Canagliflozin 300 mg (N=84) | Canagliflozin 300 mg/Phentermine 15 mg (N=83)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 2 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 11 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 6 | 7 | 3
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 2 | 0
Acute Sinusitis (Infections and infestations) | 2 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 5 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 3 | 3
Influenza (Infections and infestations) | 1 | 4 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Pharyngitis Streptococcal (Infections and infestations) | 1 | 1 | 4 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 2 | 3
Tooth Infection (Infections and infestations) | 4 | 1 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 15 | 5 | 11 | 9
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 3 | 2
Viral Infection (Infections and infestations) | 0 | 1 | 2 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 0 | 3 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 4 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 3 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 2 | 3 | 5
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 0 | 2
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.